CLINICAL TRIAL: NCT07341646
Title: The Effect of Endotracheal Tube Cuff Pressure Assessment Methods on Postoperative Complications in Patients Undergoing Elective Breast Surgery: A Randomized Controlled Trial
Brief Title: Effect of Cuff Pressure Assessment Methods on Postoperative Complications in Breast Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ahmet Salih Tüzen, MD, Medical Doctor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-KAEK-23
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Airway Complications; Postoperative Sore Throat; Hoarseness; Dysphagia; Cough Severity
Keywords: Continuous Cuff Pressure Monitoring; Manometer; Endotracheal Tube Cuff Pressure; Postoperative Sore Throat; Airway Complications; Intubation Safety
MeSH Terms: conditions — Hoarseness; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: This study utilizes a parallel-group design with a 1:1:1 allocation ratio. Participants are randomized into three distinct arms: continuous pressure monitoring, intermittent manometer measurement, and a control group utilizing the minimal occlusive volume technique. The study employs a single-blind masking protocol wherein the outcomes assessor is blinded to the intervention assignment to minimize detection bias. This model is designed to compare the efficacy of objective versus subjective cuff pressure management strategies in preventing postoperative upper airway complications within a homogenous population of elective breast surgery patients.
Who Masked: Outcomes Assessor
Masking Description: Due to the distinct physical differences between the devices and techniques used (continuous pressure indicator, manual manometer, or standard syringe), the anesthesiologist performing the intubation and cuff pressure adjustment cannot be blinded to the group assignment. However, to ensure study integrity, the outcome assessors responsible for collecting postoperative data and scoring symptoms (sore throat, hoarseness, dysphagia, etc.) at 0, 1, 12, and 24 hours will be strictly blinded to the patient's allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous Pressure Indicator Group (Experimental): Patients in this group will have their endotracheal tube cuff pressure continuously monitored and maintained within the range of 20-30 cmH₂O using a continuous pressure indicator device throughout the surgery.
  Interventions: Device: Continuous Cuff Pressure Indicator
- Manometer Group (Active Comparator): Patients in this group will have their endotracheal tube cuff pressure measured and adjusted once using a manual manometer immediately after intubation to a target range of 20-30 cmH₂O.
  Interventions: Device: Manual Cuff Pressure Manometer
- Control Group (Minimal Occlusive Volume) (Active Comparator): Patients in this group will have their endotracheal tube cuff inflated using the minimal occlusive volume technique (inflating until the air leak stops) without the use of a pressure gauge.
  Interventions: Procedure: Minimal Occlusive Volume Technique

INTERVENTIONS:
Device: Continuous Cuff Pressure Indicator — A device utilized to continuously monitor the endotracheal tube cuff pressure intraoperatively. It allows for real-time observation and maintenance of the pressure within the target range of 20-30 cmH₂O throughout the surgery.
  Other Names: Continuous Cuff Pressure Controller
  Arms: Continuous Pressure Indicator Group
Device: Manual Cuff Pressure Manometer — A standard analog manometer used for a single-time measurement of the endotracheal tube cuff pressure immediately after intubation. The pressure is adjusted to the standard range of 20-30 cmH₂O and not monitored continuously thereafter.
  Other Names: Handheld Cuff Manometer
  Arms: Manometer Group
Procedure: Minimal Occlusive Volume Technique — A standard clinical technique where the endotracheal tube cuff is inflated with the minimum volume of air required to prevent audible air leakage during positive pressure ventilation. No objective pressure gauge is used for adjustment.
  Other Names: Leak Test Method
  Arms: Control Group (Minimal Occlusive Volume)

SUMMARY:
Endotracheal intubation is a standard procedure used to secure the airway during general anesthesia. A key component of the breathing tube is the "cuff," a balloon-like device that is inflated to seal the airway and prevent aspiration. However, if the pressure within this cuff is too high, it can restrict blood flow to the tracheal lining, leading to complications such as postoperative sore throat, hoarseness, and difficulty swallowing (dysphagia).

Currently, there are various methods to monitor and adjust this pressure. In many clinical practices, the pressure is adjusted subjectively or checked only once at the beginning of the surgery. These methods may allow pressure to exceed safe limits (typically 20-30 cmH₂O) or fluctuate during the procedure, potentially causing tissue irritation. This randomized controlled trial aims to compare three different methods of assessing and maintaining endotracheal tube cuff pressure to determine which is most effective at reducing postoperative complications. The study focuses on women undergoing elective breast surgery, a group chosen because the surgery typically lasts 1-3 hours and does not involve major changes in head and neck position, allowing for a clear assessment of the cuff pressure methods.

Participants will be randomly assigned to one of three groups:

* Continuous Monitoring Group: Cuff pressure is monitored continuously using a pressure indicator and maintained within the 20-30 cmH₂O range throughout the surgery.
* Manometer Group: Cuff pressure is measured and set to 20-30 cmH₂O using a manual manometer once, immediately after intubation.
* Control Group (Minimal Occlusive Volume): The cuff is inflated with the minimum amount of air required to prevent an air leak, without using a pressure gauge.

Researchers will assess patients for sore throat, cough, hoarseness, and swallowing difficulties at 0, 1, 12, and 24 hours after surgery to identify the safest and most comfortable method for airway management.

DETAILED DESCRIPTION:
This prospective, randomized, parallel-group, single-blind clinical trial investigates the efficacy of different endotracheal tube cuff pressure monitoring techniques in preventing postoperative airway morbidity. The study will be conducted at the İzmir Kâtip Çelebi University Atatürk Training and Research Hospital, Department of Anesthesiology and Reanimation.

The study population consists of female patients aged 18-65 years, classified as ASA I-III, who are scheduled for elective breast surgery under general anesthesia requiring endotracheal intubation. Breast surgery patients were selected as the target population because they represent a homogenous group (typically healthy females), undergo procedures of moderate duration (1-3 hours), and remain in a fixed supine position without significant head-neck manipulation, thereby minimizing confounding variables that could affect cuff pressure.

Study Procedures and Randomization: A total of 90 eligible patients will be enrolled. After providing informed consent, participants will be randomized into three groups with a 1:1:1 allocation ratio. Randomization will be performed using a computer-generated random sequence (via Research Randomizer, randomizer.org) to ensure unbiased assignment. The allocation sequence will be concealed from the investigators until the patient has been successfully intubated.

The three study arms are defined as follows:

* Continuous Pressure Indicator Group: Cuff pressure will be continuously monitored and maintained within the therapeutic range of 20-30 cmH₂O using a continuous pressure indicator device throughout the surgery.
* Manometer Group: Following intubation, the cuff pressure will be measured once using a manual manometer and adjusted to the 20-30 cmH₂O range. No further adjustments will be made unless clinically indicated.
* Control Group (Minimal Occlusive Volume): The cuff will be inflated using the "minimal occlusive volume" technique, wherein the cuff is inflated with the minimum volume of air required to prevent audible air leaks. No objective pressure gauge will be used.

Anesthesia Protocol: All patients will receive a standardized anesthesia protocol. Induction will be achieved with appropriate intravenous agents, and intubation will be performed by the same experienced anesthesiologist to ensure consistency. Anesthesia maintenance will be uniform across all groups. The study excludes patients with a history of difficult intubation, recent respiratory tract infections (within 6 months), preoperative sore throat/hoarseness, or operative times exceeding 3 hours.

Data Collection and Outcomes: The primary outcome is the incidence and severity of postoperative sore throat. Secondary outcomes include hoarseness, cough, dysphagia, laringospasm/bronchospasm, hemorrhage, and recovery times (extubation time, time to spontaneous respiration, and PACU stay duration).

Outcomes will be assessed at four specific time points:

* 0 hours (immediately post-extubation)
* 1 hour (in the Post-Anesthesia Care Unit - PACU)
* 12 hours (on the ward)
* 24 hours (postoperative day 1)

A four-point scale (0-3) will be used to grade symptoms (e.g., 0=None, 1=Mild, 2=Moderate, 3=Severe). To ensure blinding, the postoperative symptom assessment will be performed by a researcher who is unaware of the patient's group assignment.

Statistical Analysis: Sample size calculation indicated that 81 patients are required to detect a significant difference (effect size f=0.41, power=0.90, alpha=0.05), which was increased to 90 to account for a 10% dropout rate. Data will be analyzed using SPSS 26.0. Continuous variables will be analyzed using ANOVA or Kruskal-Wallis tests depending on normality, and categorical variables will be analyzed using Chi-square or Fisher's exact tests. Repeated measures (time-dependent changes) will be analyzed using the Friedman test.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 65 years.
* Patients classified as American Society of Anesthesiologists (ASA) physical status I, II, or III.
* Patients scheduled for elective breast surgery requiring general anesthesia and endotracheal intubation.
* Patients who provide voluntary written informed consent to participate.

Exclusion Criteria:

* Patients with a history of Chronic Obstructive Pulmonary Disease (COPD) or an asthma attack within the last 6 months.
* Presence of preoperative sore throat, hoarseness, or cough.
* Patients with predicted difficult intubation or those who are difficult to intubate.
* Patients with communication difficulties that prevent accurate assessment of symptoms.
* Patients whose surgery duration exceeds 3 hours.
* Patients older than 65 years.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Postoperative Sore Throat | 4 time points: Baseline (post-extubation), 1st, 12th and 24th hour following extubation.
  Postoperative sore throat will be assessed using a 4-point categorical scale. The scoring is defined as follows: 0 = No sore throat; 1 = Mild sore throat (less than a cold); 2 = Moderate sore throat (similar to a cold); 3 = Severe sore throat (worse than a cold). Higher scores indicate a more severe adverse outcome.

SECONDARY OUTCOMES:
Incidence and Severity of Hoarseness | 4 time points: Baseline (post-extubation), 1st, 12th and 24th hour following extubation.
  Assessed using a 4-point scale: 0 = None; 1 = Mild (minimal change in speech); 2 = Moderate (obvious hoarseness, communication not affected); 3 = Severe (affects communication)
Incidence and Severity of Cough | 4 time points: Baseline (post-extubation), 1st, 12th and 24th hour following extubation.
  Assessed using a 4-point scale: 0 = None; 1 = Mild (occasional); 2 = Moderate (frequent, disturbing); 3 = Severe (uncontrolled, constant, painful).
Incidence and Severity of Dysphagia | 4 time points: Baseline (post-extubation), 1st, 12th and 24th hour following extubation.
  Difficulty swallowing assessed using a 4-point scale: 0 = None; 1 = Mild (mild difficulty with solid foods); 2 = Moderate (obvious difficulty with solids and liquids); 3 = Severe (limits oral intake).
Incidence of Laryngospasm or Bronchospasm | Up to 30 minutes following extubation.
  The presence (Yes) or absence (No) of laryngospasm or bronchospasm occurring during the extubation phase.
Incidence of Airway Hemorrhage | At the time of extubation
  Presence of blood on the endotracheal tube or in the airway immediately following extubation (Yes/No).
Extubation Time | Up to 30 minutes following surgery completion.
  The duration in minutes from the completion of the surgery to the removal of the endotracheal tube.
Time to Spontaneous Respiration | Up to 30 minutes following extubation.
  The time in minutes from the discontinuation of anesthetic agents to the return of adequate spontaneous ventilation.
Early Recovery Time | Up to 30 minutes following extubation.
  The time in minutes from extubation to the achievement of recovery criteria on the operating table (responding to verbal stimuli, head lift for 5 seconds, swallowing) prior to PACU transfer.
Duration of Post-Anesthesia Care Unit (PACU) Stay | Up to 24 hours following extubation.
  The total duration in minutes the patient remains in the recovery room until discharge criteria are met.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Aksun, M.D., Principal Investigator — Izmir Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Izmir Katip Celebi University Atatürk Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data necessary to support the study protocol, including de-identified individual participant data (IPD) related to study protocol, and primary and secondary outcome measures, will be made available upon reasonable request from qualified researchers for academic purposes, in accordance with institutional and ethical guidelines.

REFERENCES:
- [Result] Wang C, Yan X, Gao C, Liu S, Bao D, Zhang D, Jiang J, Wu A. Effect of continuous measurement and adjustment of endotracheal tube cuff pressure on postoperative sore throat in patients undergoing gynecological laparoscopic surgery: a randomized controlled trial. J Clin Monit Comput. 2024 Dec;38(6):1379-1386. doi: 10.1007/s10877-024-01173-y. Epub 2024 May 11. PMID 38733506
- [Result] Nwosu ADG, Ossai EN, Ejezie C, Obodo OC. Educational Intervention Can Improve the Pilot Balloon Palpation Method of Tracheal Tube Cuff Pressure Monitoring: An Experimental Study. J West Afr Coll Surg. 2025 Jan-Mar;15(1):53-58. doi: 10.4103/jwas.jwas_162_23. Epub 2024 Aug 2. PMID 39735817
- [Result] Maertens B, Blot K, Blot S. Prevention of Ventilator-Associated and Early Postoperative Pneumonia Through Tapered Endotracheal Tube Cuffs: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Crit Care Med. 2018 Feb;46(2):316-323. doi: 10.1097/CCM.0000000000002889. PMID 29206767
- [Result] Vasanth Karthik R, Ranganathan P, Kulkarni AP, Sharma KS. Does cuff pressure monitoring reduce postoperative pharyngolaryngeal adverse events after LMA-ProSeal insertion? A parallel group randomised trial. J Anesth. 2014 Oct;28(5):662-7. doi: 10.1007/s00540-014-1811-0. Epub 2014 Mar 19. PMID 24643810
- [Result] Choi HR, Kim S, Kim HJ, Ahn EJ, Kim KW, Bang SR. [Endotracheal tube cuff pressure increases in patients undergoing shoulder arthroscopy: a single cohort study]. Braz J Anesthesiol. 2020 Nov-Dec;70(6):583-587. doi: 10.1016/j.bjan.2020.04.021. Epub 2020 Nov 18. PMID 33279230
- [Result] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989